CLINICAL TRIAL: NCT03564223
Title: The Great Ormond Street Hospital Top Child and Adolescent Health Study
Status: Completed | Type: Observational
Sponsor: Institute of Child Health (Other)
Responsible Party: Sponsor
Other Study IDs: 18DD02; IRAS Project ID: 238932 (Other: Health Research Authority (HRA), United Kingdom)
Record Dates: First submitted 2018-06-11; First posted 2018-06-20 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Adolescent Behavior; Child Behavior; Parents
Keywords: Adolescent; Parental concerns; Child Health; Paediatrician Concerns
MeSH Terms: conditions — Adolescent Behavior; Child Behavior

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parents/Guardians: Parents/Guardians aged over 18, attending Great Ormond Street Hospital Outpatients.
  Intervention: Administer questionnaire to review and decide on significance of each of 30 child health concerns
- Paediatricians: Paediatricians working at Great Ormond Street Hospital NHS Foundation Trust.
  Intervention: Administer questionnaire to review and decide on significance of each of 30 child health concerns

SUMMARY:
The Great Ormond Street Hospital (GOSH) Top child and adolescent health problems study aims to identify the top health concerns that parents/guardians and paediatricians in a tertiary hospital have for young people in England. 400 parents or guardians attending GOSH outpatients and 200 Paediatricians working at GOSH will be asked to rank a list of 30 child health concerns and results compared. Analysis will be done by demographics as well.

DETAILED DESCRIPTION:
The GOSH top child and adolescent health problems study aims to identify the top health concerns that parents/guardians and paediatricians in a tertiary hospital have for young people in England. The study will be surveying parents/guardians and paediatricians at Great Ormond Street Hospital (GOSH), asking them to review and give their impressions from a list of thirty common child and adolescent health issues. Analysis of responses will provide a list of problems that are most important and determine if respondents feel that the NHS England is adequately addressing these problems.

The project was designed with public partnership. The investigators conducted literature reviews, and adopted with permission, a survey instrument used by the C.S. Mott Children's Hospital National Poll in Michigan, USA. Some parents were asked to list child and adolescent health problems that they deemed most important. A consensus meeting with experts was held, to select the thirty most common and important public health issues for young people in England, from which the study will identify problems with the highest concern. This project and its intended outcomes will span medical, nursing, research and voluntary services that will improve child and adolescent healthcare provision the UK.

The State of Child Health (SoCH) Report 2017 highlights indicators of child health problems across the four nations of the United Kingdom. There are some polls that were conducted in Australia and USA, investigating the top concerns for child health problems and thus providing a framework onto which to find solutions. The Royal Children's Hospital Melbourne through its National Child Health Poll established that that excessive screen time was the greatest parental concern, and that the top ten concerns related to modern lifestyle, mental health and child safety. Similarly, the C.S. Mott Children's Hospital National Poll on children's health selected a national sample of adults to identify health topics that are a "big problem" for children and teenagers. The 2017 report identified bullying/cyberbullying as the greatest concern. However there is no available evidence about studies being conducted in the United Kingdom to find out what parents/guardians and paediatricians report as the top child and adolescent health problems.

The information would be valuable to the health professionals at the point of care, as well as the national healthcare system. This study analyses information from groups on both the supply and demand side of child and adolescent healthcare. Understanding the different perceptions of child and adolescent health problems between healthcare professionals and parents/guardians can lead to improved follow-up care and compliance with advice. Information from this study can be used as a basis for the establishment of a UK national poll that would further investigate public concerns for child health.

ELIGIBILITY:
Inclusion Criteria:

* Parents/Guardians attending GOSH NHS Foundation Trust Outpatients
* Paediatricians practicing at GOSH

Exclusion Criteria:

* Parents/Guardians and Paediatricians outside the GOSH or NHS England
* Children aged under 18 years old
* Inpatients
* Parents/Guardians who cannot communicate in English and do not have an interpreter
* Participants who have previously responded to the questionnaire
* Outpatient coordinator or Nurse in Charge feels that the potential participant may be vulnerable, or have complex issues.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Parents/guardians attending GOSH OPD (nA)
  * Target Population = Yearly OPD attendance = 308,457
  * Confidence Level is 95%
  * Margin of error = 5%
  * Target Sample Size = 384, approximately 400
  * Sampling will be matched to attendance proportions in the six OPD areas - Cheetah, Manta ray, Rhino, Zebra, Hare and Hippo.
  Paediatricians (nB)
  * Target population = 400 Paediatricians at GOSH
  * Confidence Level is 95%
  * Margin of error = 5%
  * Target Sample Size = 197, approximately 200
  * There will be no power calculation done. No statistical testing will be conducted
Sampling Method: Non-Probability Sample
Enrollment: 425 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-06-28 (Actual)

PRIMARY OUTCOMES:
Determination of Top 10 Child Health Concerns | 12 Months
  Ranking of Top Child Health Concerns by Parents and Paediatricians, which will obtained by asking both groups to state on a 4-point Likert scale on how they rate the significance of each of 30 child health concerns.
  4 categorical ordinal responses from better to worse; Not a problem, small problem, moderate problem and large problem. These rankings will be analysed with weighted values assigned (0, 1, 2, 3). There is an option for I don't know.
  This will enable determination of top 10 child health concerns
Adequacy of NHS perceptions | 12 Months
  Parents and Paediatricians are asked to decide if they think the NHS is adequately addressing adolescent and child health issues, on a 5-point Likert scale rating agreement with the statement.
  5 categorical ordinal responses from better to worse; Strongly agree, agree, neutral, disagree, strongly disagree. These rankings will be recoded in analysis as 'Disagree' (Strongly disagree, disagree) and 'Do not disagree' (Neutral, agree, strongly agree).
Determination of Top 3 information sources for parents and paediatricians | 12 Months
  Parents and Paediatricians are asked to list their top three information sources, and these will be analysed to determine the three most common sources of information for each group.

CONTACTS AND LOCATIONS:
Overall Officials: Vikram Palit, Principal Investigator — Great Ormond Street Hospital Institute of Child Health
Locations (1):
- Great Ormond Street Institute of Child Health, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There is currently no plan made to share IPD. This project is part of an educational project for the fulfillment of an MSc. Paediatrics and Child Health at University College London.

REFERENCES:
- [Result] Garbutt JM, Leege E, Sterkel R, Gentry S, Wallendorf M, Strunk RC. What are parents worried about? Health problems and health concerns for children. Clin Pediatr (Phila). 2012 Sep;51(9):840-7. doi: 10.1177/0009922812455093. Epub 2012 Jul 26. PMID 22843294
- See also: C.S. Mott Poll for Top Child Health Concerns — https://mottpoll.org/tags/top-10-child-health-concerns
- See also: Royal Children's Hospital Melbourne Child Health Poll — https://www.rchpoll.org.au/polls/top-10-child-health-problems/
- See also: State of Child Health Report 2017 — https://www.rcpch.ac.uk/resources/state-child-health-report-2017

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-04): https://cdn.clinicaltrials.gov/large-docs/23/NCT03564223/Prot_SAP_000.pdf